CLINICAL TRIAL: NCT07102082
Title: Ifluence of Authorized Smokeless Tobacco Product Modified Risk Claims II: Laboratory Assessment of Sensory and Subjective Effect
Brief Title: Influence of Authorized Smokeless Tobacco Product Modified Risk Claims I: Consumer Product Demand
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I-4008824; R21CA289541 (NIH)
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Smoking Behaviors
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A - no claim (Sham Comparator): Participants view smokeless tobacco ads with no claims
  Interventions: Behavioral: Modified Risk - None
- Group B - Modified Risk Tobacco Product Claim (Active Comparator): Participants view ads with a modified risk claim
  Interventions: Behavioral: Modified Risk Claim

INTERVENTIONS:
Behavioral: Modified Risk - None — Participants view ads with no modified risk claim
  Arms: Group A - no claim
Behavioral: Modified Risk Claim — Participants view ads with a modified risk claim
  Arms: Group B - Modified Risk Tobacco Product Claim

SUMMARY:
To explore consumer responses to the announcement and implementation of new modified risk claims for Copenhagen and General Snus (brands of smokeless tobacco (ST) products) using a series of complementary and innovative research activities and methods.

DETAILED DESCRIPTION:
Primary Objectives:

To assess the influence of smokeless tobacco products' modified risk claims on:

1. Product demand (measured as willingness to pay in USD) using an experimental auction approach; and
2. Perceived risk of tobacco-associated diseases as assessed using questionnaire-based measures.

ELIGIBILITY:
Inclusion Criteria:

* Residing in one of the 8 counties of Western New York (Erie, Niagara, Cattaraugus, Chautauqua, Allegheny, Livingston, Genesee, Orleans, Wyoming).
* Smoke cigarettes every day, at least 5 cigarettes per day, for at least 1 year.
* Open to trying a non-combusted oral tobacco product.
* Have access to a device (ie: computer/tablet/smartphone) with internet capabilities to participate in an online survey study.
* Have the ability to read, write, and communicate in English.
* Participant must understand the investigational nature of this study and an Independent Ethics Committee/Institutional Review Board approved information sheet prior to receiving any study related procedure

Exclusion Criteria:

* Plan to quit smoking in the next 30 days.
* Use of smokeless tobacco at least weekly in the last 6 months.
* Lifetime use (that is, ever used at any time prior to the study) of Copenhagen or General Snus.
* Unwilling or unable to follow protocol requirements.
* Pregnant or planning to become pregnant (by self report)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Demand for cigarettes | After one session - 1 hour
  After watching a series of advertisements for oral smokeless tobacco products, participants will provide opinions of them, including likelihood of buying product.
Increase in knowlege of tobacco-associated diseases | After one session - I hour
  multi item assessment questionnaires of perceived harm/risks from products

CONTACTS AND LOCATIONS:
Overall Officials: Richard O'Connor, Principal Investigator — Roswell Park
Locations (1):
- Roswell Park, Buffalo, New York, United States